CLINICAL TRIAL: NCT06884748
Title: PREVENTION OF RECURRENCE OF CLOSTRIDIOIDES DIFFICILE COLITIS WITH URSODEOXYCHOLIC ACID (UCDA) AS A SUPPLEMENT TO STANDARD THERAPY
Acronym: PREVENT
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Daniel Stein, Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRO00049268
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-05

CONDITIONS: Clostridioides Difficile Infection
Keywords: Clostridioides difficile infection
MeSH Terms: conditions — Clostridium Infections | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- UDCA Arm (Experimental): Standard of care treatment (Flagyl, Vancomycin or Fidaxomicin) + UDCA 500 mg TID for 8 weeks. UDCA to be started while patient is on antibiotics for C. difficile and continue for 8 weeks total.
  Interventions: Drug: Ursodiol 500 MG

INTERVENTIONS:
Drug: Ursodiol 500 MG — Standard of care treatment (Flagyl, Vancomycin or Fidaxomicin) + UDCA 500 mg TID for 8 weeks. UDCA to be started while patient is on antibiotics for C. difficile and continue for 8 weeks total.

SUMMARY:
The goal of this clinical trial is to determine whether Ursodeoxycholic Acid (UDCA) can help prevent recurrence of Clostridioides difficile (C. diff) colitis when used along with standard antibiotic treatment. C. diff colitis is a serious infection that can return after treatment, and researchers want to see if UDCA can reduce this risk.

This study aims to answer three main questions. First, can UDCA help prevent C. diff from returning after standard treatment? Second, does adding UDCA to treatment lower the need for repeated antibiotic use? Third, is UDCA safe and well-tolerated for people with C. diff?

Participants in the study will be adults diagnosed with C. diff colitis who have risk factors for recurrence. Each participant will receive standard antibiotic treatment, which may include Vancomycin, Fidaxomicin, or Metronidazole. In addition to their antibiotic therapy, participants will take UDCA at a dose of 500 mg three times a day for up to eight weeks. If a participant's stool test shows they are C. diff negative at four weeks, they will stop taking UDCA early.

Researchers will monitor participants throughout the study. Stool samples will be tested at the beginning, after four weeks, and at the end of the study. If a participant develops diarrhea, a stool test will check for C. diff. If C. diff is negative, the UDCA dose will be reduced. Weekly phone calls will be made to check for side effects and ensure participants are following the treatment plan.

C. diff colitis is a common and serious infection, with up to 46 percent of high-risk patients experiencing recurrence. Current treatments rely on antibiotics, which can disrupt gut bacteria and increase the risk of reinfection. UDCA is a naturally occurring bile acid that may help prevent C. diff from growing, reducing the need for repeated antibiotic treatment. If successful, this study could introduce a new way to prevent C. diff from coming back, helping patients recover more effectively while reducing antibiotic use.

Eligible participants must be at least 18 years old, have a positive C. diff test, and be receiving standard antibiotic treatment for C. diff. People who have severe or life-threatening C. diff colitis, a life expectancy of less than six months, serious liver disease, or are pregnant or breastfeeding will not be eligible to participate.

UDCA is FDA-approved and has been used safely for decades in liver diseases and gallstone treatment. Some people may experience mild side effects, such as diarrhea, nausea, or stomach discomfort. Participants will be closely monitored for safety throughout the study.

This trial will take place within the Froedtert and Medical College of Wisconsin healthcare system in Milwaukee, Wisconsin.

DETAILED DESCRIPTION:
Prevention of Recurrence of Clostridioides Difficile Colitis with

Ursodeoxycholic Acid (UCDA) as a Supplement to Standard Therapy

Paraj D. Patel M.D, Daniel J. Stein, M.D, Helmut V. Ammon, MD

This proposal describes the use of UDCA as an adjunct to standard treatment of C. difficile (C. diff) colitis for the prevention of recurrence of the disease.

The Problem: C. diff colitis is a serious burden on the healthcare system. In 2011 there were close to 500,000 cases of and 29,000 deaths from C. diff. colitis reported in the US at an annual cost of 58 billion dollars [1, 2] Treatment consists of Vancomycin or Fidaxomicin [3]. The recurrence rate is between 7% and 20% within 2 months [1, 4]. The risk of recurrence increases with each episode and various risk factors to up to 46% in the presence of more than 3 risk factors[5, 6]. Current efforts to deal with this problem include prolonged treatment with antibiotics, fecal microbiota transplants, probiotics, and monoclonal antibodies [7] .

Recurrent C. diff. infection is associated with is a loss of diversity in the fecal microbiome and the consequent loss of the ability to deconjugate bile acids [6, 8]. Stool from patients with recurrent C. diff. colitis requiring fecal transplant contains mainly taurocholate and no secondary bile acids [9]. In in vitro studies taurocholate facilitates the germination of C. difficile spores and the growth of the vegetative form [10]. For this reason, taurocholate is used in the growth medium for the culture of C. diff [9]. Treatment of recurrent C. diff. colitis with fecal transplants is directed at restoration of the diversity of the fecal microbiome and restoration of a normal fecal bile acid profile [3, 11, 12]

The Solution:

UDCA, a secondary bile acid derived from chenodeoxycholic acid in the human colon, inhibits the germination of C. diff in vitro at a and its growth of the vegetative form in concentration as low as 0.5 mmol/L [13, 14]

This observation prompted the use of UDCA (1200 mg/day) for the successful treatment of a patient with an ileo-anal pouch with recurrent intractable C. difficile pouchitis [14]. A subsequent uncontrolled case series reported the successful control of recurrent C. difficile colitis in 14 out of 16 patients with UDCA (600 - 900 mg/day) given for 29 - 235 days[15].

Three different studies using different experimental designs indicate that UDCA is poorly absorbed and that adequate doses of UDCA could deliver adequate colonic concentrations to prevent germination and inhibit growth of C. difficile [16-18]

Experimental Design and Calculation of Sample size

We assume that a higher dose of UDCA (1500 mg/day) could improve the results observed by Webb et al [15]. Assuming a fecal weight of 400g/day (diarrhea) with the corresponding volume of distribution of 400 ml the patients in the study by Webb et al [14] would have had a fecal concentration of UDCA of 1.8 mmol/L, based on the absorption rates observed by Walker et al [17]. The dose of UDCA in our proposal (1500 mg/day) would result in a fecal UDCA concentration of 7 mmol/L, well above the 0.5 mmol/l inhibiting vegetative growth of C. diff in vitro [11,12]

For the exploratory study we propose to use a single arm, open label design with historical controls. Use of historical controls is justified if the study population is small, as in our single center study, and the outcome in question is dichotomous [19].

As historical controls we will use the placebo group of the treatment trial of the use of Bezlutoxumab for the prevention of the recurrence of C. difficile colitis [7]. Using patients with ≥1 risk factors we would get a sample size in the control group of n = 468 with a recurrence rate of 37.2 %. Since the outcome is dichotomous (Recurrence yes/no) we used the ClinCalc sample size calculator to determine the necessary Number to Treat. Assuming a 12.5% recurrence rate for a minimal response [13] the necessary Number to Treat is 25 (plus 2 to account for drop-outs) (for Type I/II error: Alpha 0.05; Beta 0.2; Power 0.8). In the study the proposed dose of UDCA will be 1500 mg/day (approximately 20 mg/kg/day) in divided doses. The dose was chosen to get adequate colonic concentrations of UDCA while reducing the risk of drug induced diarrhea [18-22]. The duration of treatment will be 60 days, the time interval for most recurrences to occur [1, 3].

Safety:

UDCA has been widely used for the dissolution of gallstones prior to the advent of laparoscopic cholecystectomy [20] and is currently the FDA approved treatment of choice for Primary Biliary Cholangitis (PBC)[21]. It is the treatment of choice for cholestasis of pregnancy (ICP)[22], and for the prevention of gallstone formation after gastric bypass surgery [23]. It is also being used for treatment of primary sclerosing cholangitis (PSC) [24], liver disease due to cystic fibrosis [25], and for the prevention of hepatic complications in allogenic stem cell transplantation [26].

The safety of the administration of UDCA as high as 30 mg/kg/24 hours (50 % higher than in our proposal) is well established. Nine studies report the use of UCDA 28-35 mg/kg/day for weeks to 3 years in treatment trials in 378 patients, 74 with PBC [27, 28], 115 with PSC [29-31], 169 with nonalcoholic steato-hepatitis (NASH)[32-34], and 20 with ICP [22]

Only one study of patients with NASH reports significant side effects (diarrhea in 38.7% vs. 17.2 % in the placebo group (p<0.01) and abdominal discomfort in 25.8% vs. 10.9% (p<0.04) [34]. One study of 12 patients with NASH reported diarrhea in 2 and fatigue and pruritus in 1 [33]. One study of 54 patients with PBC reports 2 cases with diarrhea, 2 with nausea and vomiting, 1 with thrombocytopenia, and 1 with a skin rash [27]. In a study of patients with NASH 11/95 patients receiving UDCA developed diarrhea vs 1/91 in the placebo group [32]. In a study of 10 patients with PSC receiving high dose UDCA one developed cholangitis, 1 underwent cholecystectomy and 1 reported loss of libido [29]. The largest study of the use of high dose UDCA in PSC was terminated after three years because of a higher incidence of adverse effect on outcomes of the liver disease in comparison to the placebo group [31]. A retrospective analysis of this study also found a higher incidence of neoplastic changes in the colon in patients with chronic ulcerative colitis in comparison with the control group after 2 years of therapy [35]. Taking all studies together 17.9 % of patients receiving high dose UDCA developed diarrhea. A systematic review of the literature found no serious side effects with the use of UDCA [36]

We therefore feel justified to test the ability of UDCA administered at a dose of 1500 mg/day in divided doses (approximately 20 mg/kg/day) to prevent the recurrence of C. difficile colitis in a pilot program, enrolling consecutive patients and comparing the outcome to historical controls.

PROTOCOL

.

Eligible patients: C. diff. toxin +ve patients > 18 years with one or more risk factors for recurrence [6,7] requiring standard treatment with Flagyl, Vancomycin or fidaxomicin.

Exclusion criteria: Life expectancy < 6 months; fulminant colitis; ileus; decompensated liver disease; pregnancy and lactating females; Inability to give informed consent.

Treatment: Standard treatment (Flagyl, Vancomycin or Fidaxomicin) + UDCA 500 mg TID. UDCA to be started while patient is on antibiotics for C. diff. for 8 weeks (unless C. diff negative by 4 weeks).

Follow-up for 6 moths.

Endpoint: Relapse yes/no

Monitoring:

Check stool for C. diff (PCR/toxin) at entry, at 4 weeks, and at completion. If C. diff negative by 4 weeks stop treatment. If patient reports diarrhea, check stool for C. diff. toxin. If negative, reduce UDCA by 25%.

Weekly telephone call to patient to check on side effects and encourage compliance

Ribotyping of C. diff at entry

Recruitment:

Potential patient pool: Patients within the Froedtert/MCW health care

system in the greater Milwaukee area

Lab issues daily list of C. diff positive patients

Obtain permission from PCP to contact patient,

Screen for exclusions,

Obtain informed consent,

Enroll patient,

Budget:

Number of patients: 27

Medication: Ursodeoxycholic acid 500 mg capsules: (n=4,860)

Pharmacy quote: $ 96.78/100 $ 4,704.--

Cost of stool test for C. difficile at 4 and 8 weeks

Cost for profiling of C. diff strains (ribotyping)

References

1. Lessa, F.C., et al., Burden of Clostridium difficile infection in the United States. N Engl J Med, 2015. 372(9): p. 825-34.
2. Depestel, D.D. and D.M. Aronoff, Epidemiology of Clostridium difficile infection. J Pharm Pract, 2013. 26(5): p. 464-75.
3. Surowiec, D., et al., Past, present, and future therapies for Clostridium difficile-associated disease. Ann Pharmacother, 2006. 40(12): p. 2155-63.
4. Liu, C., et al., Insights into the Evolving Epidemiology of Clostridioides difficile Infection and Treatment: A Global Perspective. Antibiotics (Basel), 2023. 12(7).
5. Brown, K.A., et al., Meta-analysis of antibiotics and the risk of community-associated Clostridium difficile infection. Antimicrob Agents Chemother, 2013. 57(5): p. 2326-32.
6. Chang, J.Y., et al., Decreased diversity of the fecal Microbiome in recurrent Clostridium difficile-associated diarrhea. J Infect Dis, 2008. 197(3): p. 435-8.
7. Gerding, D.N., et al., Bezlotoxumab for Prevention of Recurrent Clostridium difficile Infection in Patients at Increased Risk for Recurrence. Clin Infect Dis, 2018. 67(5): p. 649-656.
8. Hofmann, A.F. and L.R. Hagey, Key discoveries in bile acid chemistry and biology and their clinical applications: history of the last eight decades. J Lipid Res, 2014. 55(8): p. 1553-95.
9. Weingarden, A.R., et al., Changes in Colonic Bile Acid Composition following Fecal Microbiota Transplantation Are Sufficient to Control Clostridium difficile Germination and Growth. PLoS One, 2016. 11(1): p. e0147210.
10. Abt, M.C., P.T. McKenney, and E.G. Pamer, Clostridium difficile colitis: pathogenesis and host defence. Nat Rev Microbiol, 2016. 14(10): p. 609-20.
11. Papazyan, R., et al., Human Fecal Bile Acid Analysis after Investigational Microbiota-Based Live Biotherapeutic Delivery for Recurrent Clostridioides difficile Infection. Microorganisms, 2023. 11(1).
12. Weingarden, A.R., et al., Microbiota transplantation restores normal fecal bile acid composition in recurrent Clostridium difficile infection. Am J Physiol Gastrointest Liver Physiol, 2014. 306(4): p. G310-9.
13. Sorg, J.A. and A.L. Sonenshein, Inhibiting the initiation of Clostridium difficile spore germination using analogs of chenodeoxycholic acid, a bile acid. J Bacteriol, 2010. 192(19): p. 4983-90.
14. Weingarden, A.R., et al., Ursodeoxycholic Acid Inhibits Clostridium difficile Spore Germination and Vegetative Growth, and Prevents the Recurrence of Ileal Pouchitis Associated With the Infection. J Clin Gastroenterol, 2016. 50(8): p. 624-30.
15. Webb, B.J., et al., Repurposing an Old Drug for a New Epidemic: Ursodeoxycholic Acid to Prevent Recurrent Clostridioides difficile Infection. Clin Infect Dis, 2019. 68(3): p. 498-500.
16. Stiehl, A., R. Raedsch, and G. Rudolph, Ileal excretion of bile acids: comparison with biliary bile composition and effect of ursodeoxycholic acid treatment. Gastroenterology, 1988. 94(5 Pt 1): p. 1201-6.
17. Walker, S., et al., Intestinal absorption of ursodeoxycholic acid in patients with extrahepatic biliary obstruction and bile drainage. Gastroenterology, 1992. 102(3): p. 810-5.
18. Invernizzi, P., et al., Differences in the metabolism and disposition of ursodeoxycholic acid and of its taurine-conjugated species in patients with primary biliary cirrhosis. Hepatology, 1999. 29(2): p. 320-7.
19. Evans, S.R., Clinical trial structures. J Exp Stroke Transl Med, 2010. 3(1): p. 8-18.
20. Bachrach, W.H. and A.F. Hofmann, Ursodeoxycholic acid in the treatment of cholesterol cholelithiasis. part I. Dig Dis Sci, 1982. 27(8): p. 737-61.
21. Lindor, K.D., et al., Primary Biliary Cholangitis: 2018 Practice Guidance from the American Association for the Study of Liver Diseases. Hepatology, 2019. 69(1): p. 394-419.
22. Mazzella, G., et al., Ursodeoxycholic acid administration in patients with cholestasis of pregnancy: effects on primary bile acids in babies and mothers. Hepatology, 2001. 33(3): p. 504-8.
23. Haal, S., et al., Ursodeoxycholic acid for the prevention of symptomatic gallstone disease after bariatric surgery (UPGRADE): a multicentre, double-blind, randomised, placebo-controlled superiority trial. Lancet Gastroenterol Hepatol, 2021. 6(12): p. 993-1001.
24. Lindor, K.D., et al., ACG Clinical Guideline: Primary Sclerosing Cholangitis. Am J Gastroenterol, 2015. 110(5): p. 646-59; quiz 660.
25. Cheng, K., D. Ashby, and R.L. Smyth, Ursodeoxycholic acid for cystic fibrosis-related liver disease. Cochrane Database Syst Rev, 2014(12): p. CD000222.
26. Ruutu, T., et al., Improved survival with ursodeoxycholic acid prophylaxis in allogeneic stem cell transplantation: long-term follow-up of a randomized study. Biol Blood Marrow Transplant, 2014. 20(1): p. 135-8.
27. Angulo, P., et al., Comparison of three doses of ursodeoxycholic acid in the treatment of primary biliary cirrhosis: a randomized trial. J Hepatol, 1999. 30(5): p. 830-5.
28. Roda, E., et al., Improved liver tests and greater biliary enrichment with high dose ursodeoxycholic acid in early stage primary biliary cirrhosis. Dig Liver Dis, 2002. 34(7): p. 523-7.
29. Cullen, S.N., et al., High dose ursodeoxycholic acid for the treatment of primary sclerosing cholangitis is safe and effective. J Hepatol, 2008. 48(5): p. 792-800.
30. Harnois, D.M., et al., High-dose ursodeoxycholic acid as a therapy for patients with primary sclerosing cholangitis. Am J Gastroenterol, 2001. 96(5): p. 1558-62.
31. Lindor, K.D., et al., High-dose ursodeoxycholic acid for the treatment of primary sclerosing cholangitis. Hepatology, 2009. 50(3): p. 808-14.
32. Leuschner, U.F., et al., High-dose ursodeoxycholic acid therapy for nonalcoholic steatohepatitis: a double-blind, randomized, placebo-controlled trial. Hepatology, 2010. 52(2): p. 472-9.
33. Adams, L.A., et al., A pilot trial of high-dose ursodeoxycholic acid in nonalcoholic steatohepatitis. Hepatol Int, 2010. 4(3): p. 628-33.
34. Ratziu, V., et al., A randomized controlled trial of high-dose ursodesoxycholic acid for nonalcoholic steatohepatitis. J Hepatol, 2011. 54(5): p. 1011-9.
35. Eaton, J.E., et al., High-dose ursodeoxycholic acid is associated with the development of colorectal neoplasia in patients with ulcerative colitis and primary sclerosing cholangitis. Am J Gastroenterol, 2011. 106(9): p. 1638-45.
36. Hempfling, W., K. Dilger, and U. Beuers, Systematic review: ursodeoxycholic acid--adverse effects and drug interactions. Aliment Pharmacol Ther, 2003. 18(10): p. 963-72.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients: C. diff. toxin +ve patients > 18 years with one or more risk factors for recurrence [6,7] requiring standard treatment with Flagyl, Vancomycin or fidaxomicin.

Exclusion Criteria:

* Life expectancy < 6 months; fulminant colitis; ileus; decompensated liver disease; pregnancy and lactating females; Inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Lack of recurrent C. difficile recurrence | 8 weeks and 3 months
  Absence of recurrent C. difficile recurrence based on symptoms and standard of care testing at 3 months and repeat stool testing at 8 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Daniel Stein, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
De Identified participant information and results
Supporting Information: Study Protocol, SAP